CLINICAL TRIAL: NCT03147196
Title: Neoadjuvant Treatment of Prostate Cancer With Bicalutamide and Raloxifene Prior to Radical Prostatectomy
Brief Title: Bicalutamide and Raloxifene Hydrochloride in Treating Patients With Prostate Cancer Undergoing Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1552; NCI-2017-00773 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1552 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Stage I Prostate Adenocarcinoma; Stage II Prostate Adenocarcinoma
MeSH Terms: interventions — bicalutamide; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (raloxifene hydrochloride) (Experimental): Patients receive low dose raloxifene hydrochloride PO daily on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Drug: Raloxifene Hydrochloride
- Arm B (bicalutamide) (Experimental): Patients receive low dose bicalutamide PO daily on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm C (raloxifene hydrochloride, bicalutamide) (Experimental): Patients receive low dose raloxifene hydrochloride PO daily and low dose bicalutamide PO on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Drug: Raloxifene Hydrochloride
- Arm D (raloxifene hydrochloride, bicalutamide) (Experimental): Patients receive high dose raloxifene hydrochloride PO daily and high dose bicalutamide PO on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Drug: Raloxifene Hydrochloride

INTERVENTIONS:
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
  Arms: Arm B (bicalutamide); Arm C (raloxifene hydrochloride, bicalutamide); Arm D (raloxifene hydrochloride, bicalutamide)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Drug: Raloxifene Hydrochloride — Given PO
  Other Names: Evista; Keoxifene Hydrochloride; LY-156758; Optruma; Raloxifene HCl; Raloxifene.HCl
  Arms: Arm A (raloxifene hydrochloride); Arm C (raloxifene hydrochloride, bicalutamide); Arm D (raloxifene hydrochloride, bicalutamide)

SUMMARY:
This phase II pilot trial studies how well bicalutamide and raloxifene hydrochloride work in treating patients with prostate cancer undergoing surgery. Antihormone therapy, such as bicalutamide and raloxifene hydrochloride, may lessen the amount of androgens made by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect and interrogate samples in patients with prostate cancer that were diagnosed with prostate cancer and are planned for radical prostatectomy at Mayo Clinic Arizona.

SECONDARY OBJECTIVES:

I. To describe the adverse event profile and tolerance of therapy for 60 days of treatment prior to surgery.

II. To assess change in stage and/or grade of cancer and prostate specific antigen (PSA) response to neoadjuvant treatment in patients with hormone sensitive prostate cancer.

TERTIARY OBJECTIVES:

I. To evaluate specific pathways and changes when comparing biopsy specimens to prostatectomy.

II. To describe the quality of life of patients receiving hormonal therapy prior to radical prostatectomy.

OUTLINE: This is a dose-escalation study. Patients are randomized to 1 of 4 arms.

ARM A: Patients receive low dose raloxifene hydrochloride orally (PO) daily on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive low dose bicalutamide PO daily on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive low dose raloxifene hydrochloride PO daily and low dose bicalutamide PO on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive high dose raloxifene hydrochloride PO daily and high dose bicalutamide PO on days 1-30. Treatment repeats every 30 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma of the prostate, >= Gleason 6, clinical stage T1a-T2c and planned for radical prostatectomy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Platelet count >= 50,000/mm^3
* Hemoglobin > 9.0 g/dL
* Creatinine =< 2.0 mg/dL
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study); Note: during the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Patients must also provide written consent for biospecimens collection on Institutional Review Board (IRB) 08-000980

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* History of a venous thromboembolic event, cerebrovascular accident (CVA), hepatic impairment, or heart failure

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Collection and interrogation of prostate cancer samples | Up to 5 years
  Pathways and biomarkers will be compared to similar analyses that have been and will be performed on in vitro and in vivo experiments. Point estimates and two-sided 95% confidence intervals will be computed.

SECONDARY OUTCOMES:
Change in cancer stage/grade via surgical pathology | Baseline up to the time of prostatectomy
  Will be calculated as the total number who were down staged divided by the number of total evaluable patients. A confidence interval for this rate will be calculated based on properties of the binomial distribution. Point estimates and two-sided 95% confidence intervals will be computed.
Incidence of adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
Percent change in PSA assessed by Prostate Cancer Clinical Trials Working Group | Baseline up to 12 weeks
  Will be calculated and displayed using waterfall plots.
Tolerance of therapy | Up to 60 days
  Proportion of patients who complete 60 days of treatment will be calculated as the number of who completed 60 days of treatment divided by the total number of evaluable patients. A confidence interval for this rate will be calculated based on properties of the binomial distribution. The proportion of patients who experience a particular event will be calculated as the total number who experienced the event of interest divided by the number of total evaluable patients, with appropriate confidence interval.

OTHER OUTCOMES:
Change in quality of life assessed using the 6-item Linear Analogue Self-Assessment and the Hormonal Domain scale of the Expanded Prostate Cancer Index Composite survey | Baseline up to 5 years
  Will be examined using stream plots and mean plots with associated two-sided 95% confidence intervals.
Change in specific pathways and biomarkers | Baseline up to 5 years
  Continuous biomarker levels will be explored in a graphical manner including mean plots and plots of change and percent change from baseline and other summary measures. Any potential relationships between the baseline level or change in the level of each biomarker and clinical outcome will be further analyzed using Wilcoxon rank sum tests or logistic regression methods, as appropriate. Association between a dichotomized biomarker and overall response will be assessed using a chi-squared test.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Castle, Principal Investigator — Mayo Clinic